CLINICAL TRIAL: NCT03321500
Title: Comparative Study of Silicone-based Soft Liner Versus Versacryl Liner for Mandibular Complete Denture Cases(Randomized Clinical Trial)
Brief Title: Measuring Quality of Life of Versacryl Relined Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Mohamed Moustafa, Internal resident at removable prosthodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: versacryl_soft liners
Record Dates: First submitted 2017-10-21; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Denture Liners

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Versacyl soft liner (Experimental): Versacryl soft liner are flexible biocompatible materials with a reported predictable long term performance, durable bonding to acrylic denture bases, high fatigue endurance, excellent wear characteristics and solvent resistance with almost no free monomer in the processed material
  Interventions: Other: Versacryl soft liner
- Silicone-based soft liner (Active Comparator): Resilient liners were introduced in the1950s and have been used since then as a gold standard material to increase the tolerance, retention and comfort of complete dentures. Resilient liners also known as 'soft liners' can be classified as temporary or permanent, cold-cured or heat-cured.Resilient liners can be divided into two main types: plasticized acrylic resins and silicone elastomers.
  Interventions: Other: Silicone-based soft liner

INTERVENTIONS:
Other: Versacryl soft liner — Versacryl has been used to construct different parts of complete and partial dentures . It can be used as thermo-elastic liner which consistency can be controlled to tailor the reline to each individual case, by adding or subtracting drops of liquid B, as explained in the directions for use. The reline can be re-adapted repeatedly, even by the patient if necessary.
  Arms: Versacyl soft liner
Other: Silicone-based soft liner — gold standard for denture relining material
  Arms: Silicone-based soft liner

SUMMARY:
Resilient liners were introduced in the1950s and have been used since then as a gold standard material to increase the tolerance, retention and comfort of complete dentures. Due to drawbacks of conventional resilient liners, their longevity is questionable and they require replacement which is time consuming and costly for the dentist and patient respectively. Versacryl is a biocompatible intraoral thermo-elastic material. So versatile, it can be used to improve esthetics, retention and comfort for the patient. It softens with heat and when it is inserted to patient's mouth, it cools to body temperature providing desired rigidity. This process can be repeated many times to ensuring the comfort for the patient. Versacryl has a reported predictable long term performance, durable bonding to acrylic denture bases, high fatigue endurance, excellent wear characteristics and solvent resistance with almost no free monomer in the processed material .

The investigators' trial is done in order to improve the longevity and oral health related quality of life of soft liners in comparison to silicone-based soft liners.

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous patients wearing complete dentures.
2. Flat mandibular residual ridge.
3. Mandibular denture indicated for relining.
4. Patients with minimum of 2 years and maximum of 5 years complete denture usage.
5. Angle's class I maxillary-mandibular relationship

Exclusion Criteria:

1. Drug or alcohol abuse.
2. Inflammatory changes in the oral cavity.
3. Candidiasis.
4. Any intra-oral soft tissue hyperplasia.
5. Physical reasons that could affect follow-up.
6. Psychiatric problems.
7. Heavy smokers.
8. Dentures indicated for remake.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
oral health related quality of life | 4 months
  OHIP-49 questionnaire

SECONDARY OUTCOMES:
tissue keratinization | 4 months
  tissue keratinization index

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krunic N, Kostic M, Petrovic M, Igic M. Oral health-related quality of life of edentulous patients after complete dentures relining. Vojnosanit Pregl. 2015 Apr;72(4):307-11. doi: 10.2298/vsp1504307k. PMID 26040175